CLINICAL TRIAL: NCT04856488
Title: Preoperative Lugol's Solution in Graves' Disease and Toxic Nodular Goiter
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Jan Calissendorff (Other)
Responsible Party: Sponsor-Investigator, Jan Calissendorff, MD, Senior Consultant, PhD, Associate Professor, Karolinska University Hospital
Organization: Karolinska University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LugolProtocol001
Record Dates: First submitted 2021-04-06; First posted 2021-04-23 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Hyperthyroidism
MeSH Terms: conditions — Hyperthyroidism | interventions — iodine potassium iodide; Solutions; Lugol's solution

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Iodine Potassium Iodide solution (Experimental): Participants receive Iodine Potassium Iodide solution oral drops 3 times per day for 10 Days prior to thyroidectomy in addition to standard preoperative treatment
  Interventions: Drug: Iodine-Potassium Iodide 5%-10% Oral and Topical Solution
- No intervention (No Intervention): Participants continue with standard preoperative treatment

INTERVENTIONS:
Drug: Iodine-Potassium Iodide 5%-10% Oral and Topical Solution — Iodine Potassium Iodide 5% oral solution, administered 3 times per day for 10 days
  Other Names: Lugol's solution
  Arms: Iodine Potassium Iodide solution

SUMMARY:
The purpose of this study is to assess if preoperative treatment with Lugol's solution prior to thyroidectomy can reduce the surgical complications hypoparathyroidism and laryngeal nerve palsy

DETAILED DESCRIPTION:
Current practice in Sweden before thyroidectomy due to hyperthyroidism is preoperative treatment with antithyroid drugs (ATD) to all patients with Graves' disease and in cases of toxic nodular goiter with pronounced hyperthyroidism. Iodine solution is administered preoperatively in selected cases of Graves' disease where ATD is intolerable. In the cases where iodine is used it is in the form of extemporaneous prepared iodine potassium iodide solution (Lugol 5%). The dose varies in clinical studies. In American and Swedish guidelines the dose is 5-10 drops 3 times per day for 10 days prior to surgery. American guidelines recommend iodine as preoperative treatment i Graves' disease but this is based on sparse evidence. Iodine as preoperative treatment in toxic nodular goiter has yet not been studied.

The purpose of this study is to assess if preoperative treatment with Lugol's solution prior to thyroidectomy due to hyperthyroidism reduce the surgical complications hypoparathyroidism and laryngeal nerve palsy.

Before including toxic nodular goiters accepted for surgery, a pilot study will be performed on 20 patients with toxic nodular goiter. They will receive Lugol solution 3 times per day for ten days and thyroid hormone levels will be measured day 0, day 3-4, day 6-7 and after 10 days of Lugol treatment. Heart rate assessed and ThyPRO39 filled out before and after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Hyperthyroidism accepted for thyroidectomy due to toxic nodular goiter with free T4 <30 pmol/L or Graves' disease
* Signed informed consent

Exclusion Criteria:

* Unstable coronary artery disease
* Previous thyroid surgery
* Congestive heart failure
* Renal insufficiency
* Hepatic failure
* Current infection
* Treatment with steroids or anticoagulants
* Thyroid associated orbitopathy CAS > 2
* Diabetes mellitus type 1
* Active cancer
* Severe psychiatric illness
* Amiodarone treatment
* Pregnancy
* Breast feeding
* Women of child bearing potential not using contraceptive
* Inability to comprehend the meaning of the study
* Iodine hypersensitivity

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 182 (Estimated)
Dates: Start 2021-11-18 (Actual); Primary Completion 2028-08 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Temporary hypoparathyroidism | 1 month postoperatively
  Numbers of participants with signs of hypoparathyroidism measured as hypocalcemia, low parathormone (PTH), supplementation with per oral vitamin D or calcium.

SECONDARY OUTCOMES:
Temporary laryngeal nerve palsy | 1 month postoperatively
  Number of patients with postoperative signs of vocal chord damage via clinical assessment or laryngoscopy.
Permanent laryngeal nerve palsy | 6 months postoperatively
  Number of patients with postoperative signs of vocal chord damage via clinical assessment or laryngoscopy.
Permanent hypoparathyroidism | 6 months postoperatively
  Numbers of participants with signs of hypoparathyroidism measured as hypocalcemia, low PTH, supplementation with per oral vitamin D or calcium.

OTHER OUTCOMES:
Change from Baseline in Quality of Life on the Thyroid Specific Patient Reported Outcome 39 (ThyPRO 29) questionnaire | 6 months postoperatively
  ThyPRO 39 is a validated thyroid specific Quality of Life form. Self reported questionnaire filled out before and after surgery. ThyPRO consists of 39 items grouped in 11 scales. Each item is is rated from 0 to 5 on a 5 point Likert scale. Increasing scores indicating decreasing quality of life. Lower scores indicating better quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Jan Calissendorff, MD, PhD, Principal Investigator — Department of Molecular Medicine and Surgery, Karolinska Institutet
Locations (1):
- Department of Endocrinology, Karolinska University Hospital, Solna, Stockholm County, Sweden

IPD SHARING:
Plan to Share IPD: Yes
The original contributions presented in the study are included in the article/supplementary material.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The original contributions presented in the study are included in the article/supplementary material. Inquiries can be directed to the corresponding author after publication.
Access Criteria: Further inquiries can be directed to the corresponding author.

REFERENCES:
- [Background] Ross DS, Burch HB, Cooper DS, Greenlee MC, Laurberg P, Maia AL, Rivkees SA, Samuels M, Sosa JA, Stan MN, Walter MA. 2016 American Thyroid Association Guidelines for Diagnosis and Management of Hyperthyroidism and Other Causes of Thyrotoxicosis. Thyroid. 2016 Oct;26(10):1343-1421. doi: 10.1089/thy.2016.0229. PMID 27521067
- [Background] Kaur S, Parr JH, Ramsay ID, Hennebry TM, Jarvis KJ, Lester E. Effect of preoperative iodine in patients with Graves' disease controlled with antithyroid drugs and thyroxine. Ann R Coll Surg Engl. 1988 May;70(3):123-7. PMID 2457351
- [Background] Randle RW, Bates MF, Long KL, Pitt SC, Schneider DF, Sippel RS. Impact of potassium iodide on thyroidectomy for Graves' disease: Implications for safety and operative difficulty. Surgery. 2018 Jan;163(1):68-72. doi: 10.1016/j.surg.2017.03.030. Epub 2017 Nov 3. PMID 29108701
- [Background] Whalen G, Sullivan M, Maranda L, Quinlan R, Larkin A. Randomized trial of a short course of preoperative potassium iodide in patients undergoing thyroidectomy for Graves' disease. Am J Surg. 2017 Apr;213(4):805-809. doi: 10.1016/j.amjsurg.2016.07.015. Epub 2016 Aug 4. PMID 27769543
- [Background] Marigold JH, Morgan AK, Earle DJ, Young AE, Croft DN. Lugol's iodine: its effect on thyroid blood flow in patients with thyrotoxicosis. Br J Surg. 1985 Jan;72(1):45-7. doi: 10.1002/bjs.1800720118. PMID 3967130
- [Background] Yilmaz Y, Kamer KE, Ureyen O, Sari E, Acar T, Karahalli O. The effect of preoperative Lugol's iodine on intraoperative bleeding in patients with hyperthyroidism. Ann Med Surg (Lond). 2016 Jun 16;9:53-7. doi: 10.1016/j.amsu.2016.06.002. eCollection 2016 Aug. PMID 27408715
- [Background] Huang SM, Liao WT, Lin CF, Sun HS, Chow NH. Effectiveness and Mechanism of Preoperative Lugol Solution for Reducing Thyroid Blood Flow in Patients with Euthyroid Graves' Disease. World J Surg. 2016 Mar;40(3):505-9. doi: 10.1007/s00268-015-3298-8. PMID 26546192
- [Background] Calissendorff J, Falhammar H. Rescue pre-operative treatment with Lugol's solution in uncontrolled Graves' disease. Endocr Connect. 2017 May;6(4):200-205. doi: 10.1530/EC-17-0025. Epub 2017 Mar 21. PMID 28325735
- [Background] Calissendorff J, Falhammar H. Lugol's solution and other iodide preparations: perspectives and research directions in Graves' disease. Endocrine. 2017 Dec;58(3):467-473. doi: 10.1007/s12020-017-1461-8. Epub 2017 Oct 26. PMID 29075974
- [Background] Spallek L, Krille L, Reiners C, Schneider R, Yamashita S, Zeeb H. Adverse effects of iodine thyroid blocking: a systematic review. Radiat Prot Dosimetry. 2012 Jul;150(3):267-77. doi: 10.1093/rpd/ncr400. Epub 2011 Oct 20. PMID 22021061
- [Background] Nauman J, Wolff J. Iodide prophylaxis in Poland after the Chernobyl reactor accident: benefits and risks. Am J Med. 1993 May;94(5):524-532. doi: 10.1016/0002-9343(93)90089-8. No abstract available. PMID 8498398
- [Derived] Hedberg F, Cramon PK, Branstrom R, Falhammar H, Calissendorff J. Assessing the impact of short-term Lugol's solution on toxic nodular thyroid disease: a pre-post-intervention study. Front Endocrinol (Lausanne). 2024 Jul 25;15:1420154. doi: 10.3389/fendo.2024.1420154. eCollection 2024. PMID 39119004